CLINICAL TRIAL: NCT05387811
Title: Characteristics and Management of Acute Kidney Injury in Hospitalized Patients With Cirrhosis: a Multicenter Intercontinental Observational Prospective Study: The International Club of Ascites GLOBAL AKI Project
Brief Title: International Registry of Acute Kidney Injury in Cirrhosis: The GLOBAL AKI Project
Acronym: GLOBAL-AKI
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera di Padova (Other)
Responsible Party: Principal Investigator, Salvatore Piano, Assistant Professor of Medicine, Azienda Ospedaliera di Padova
Other Study IDs: AOP2414
Record Dates: First submitted 2022-05-16; First posted 2022-05-24 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Liver Cirrhosis; Acute Kidney Injury; Hepatorenal Syndrome
Keywords: AKI; International Club of Ascites; Cirrhosis; Global
MeSH Terms: conditions — Liver Cirrhosis; Acute Kidney Injury; Hepatorenal Syndrome; Fibrosis | interventions — Crystalloid Solutions; Albumins; Vasoconstrictor Agents; Diuretics; Renal Replacement Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Crystalloids, albumin, vasoconstrictors, diuretics, renal replacement therapy — Adherence to International Club of Ascites recommendations for the management of AKI

SUMMARY:
The aims of this study will be to identify the clinical characteristics, the management and the outcomes of acute kidney injury in patients with cirrhosis worldwide.

Specific aims:

1. To establish the severity of AKI across different regions
2. To identify precipitants of AKI across different centers
3. To identify the phenotypes of AKI across different centers
4. To evaluate differences in the management of AKI across different centers and their impact on clinical outcomes
5. To assess outcomes of acute kidney injury (resolution of AKI, in-hospital mortality, 28-day mortality, 90-day mortality)

DETAILED DESCRIPTION:
Each center will then include patients with cirrhosis who are admitted to the hospital with AKI upon admission or who develop AKI during the hospital stay, and who provide signed informed consent.

Acute kidney injury will be defined according to the International Club of Ascites Acute Kidney Injury criteria The following precipitating events of AKI will be considered: volume loss/excessive diuretic use, spontaneous bacterial peritonitis (SBP), non-SBP infection, gastrointestinal bleeding, nephrotoxic drugs (including nonsteroidal anti-inflammatory drugs, contrast media), other causes and no identifiable precipitant.

AKI will be classified in the following phenotypes:

* Hypovolemia-induced AKI: history of excessive fluid losses (i.e., excessive diuresis due to diuretic therapy with loss of body weight >500 g/day or 1,000 g/day in patients without and with edema, respectively; severe diarrhea) or bleeding the days before AKI and improving with fluid administration.
* HRS-AKI: all the following should be present: a) ascites; b) lack of regression of AKI to a lower stage or resolution of AKI after 2 days of diuretic withdrawal and volume expansion with albumin (1 g/kg of body weight per day to a maximum of 100 g/day); c) absence of shock; d) no current or recent treatment with nephrotoxic drugs; d) absence of parenchymal disease as indicated by proteinuria >500 mg/day, microhaematuria (>50 red blood cells per high power field), urinary injury biomarkers (if available) and/or abnormal renal ultrasonography.

Patients will be followed from admission until liver transplantation, death or 90 days, whichever occurs first. Data collected will include demographic, clinical and biochemical information, such as AKI severity, phenotype and evolution. There will be particular emphasis on collecting data regarding the initial management of AKI occurring in the first 2 to 3 days. Furthermore, basic demographic and disease information will be collected in hospitalized patients with cirrhosis who do not develop AKI during the stay to determine the true burden of AKI in this patient population.

Data will be registered on an electronic case report form (eCRF) using the Research Electronic Data Capture Software REDCap.

* ATN-AKI: presence of at least three out of six of the following criteria: a) FeNa > 2%; b) urinary osmolality <400 mOsm/L; c) urinary sodium > 40 mEq/L; d) presence of shock or use of nephrotoxic drugs; e) urine sediment showing granular/epithelial casts; f) urine sediment showing renal tubular epithelial cells.
* Other parenchymal nephropathy: patients with signs of parenchymal nephropathy not qualified for a diagnosis of ATN-AKI (e.g. IgA nephropathy, glomerulonephritis, nephrotic syndrome, etc.)
* Post renal AKI: AKI caused by urinary tract obstruction (kidney/bladder stones, prostatic hyperplasia) and resolved after removal of obstruction
* Unclassified/other AKI: Other types of AKI not fulfilling the afore mentioned phenotypes

ELIGIBILITY:
Inclusion Criteria:

a) Patients with cirrhosis admitted to hospital for the treatment of a complication of liver disease (ascites, gastrointestinal bleeding, hepatic encephalopathy, bacterial infections, jaundice, etc)

Exclusion Criteria:

1. Age < 18 years old;
2. Pregnancy;
3. Hepatocellular carcinoma outside Milan criteria (i.e., a single lesion <5 cm or multiple lesions [maximum of three], the largest of which measures ≤ 3 cm);
4. Extrahepatic malignancy other than non-melanoma skin cancer within last 5 years;
5. Previously known severe extrahepatic diseases (e.g., chronic renal failure requiring hemodialysis, severe congestive heart disease [NYHA class ≥ 3]; severe chronic obstructive pulmonary disease [GOLD class ≥ 3], psychiatric disorders);
6. Previous solid organ transplantation;
7. HIV infection with CD4 ≤ 250/µL;
8. Patients who cannot provide prior informed consent and no legal surrogate decision maker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cirrhosis admitted to hospital for the treatment of a complication of liver disease (ascites, gastrointestinal bleeding, hepatic encephalopathy, bacterial infections, jaundice, etc)
  Patients without AKI will enter in a screening period during the hospitalization to identify patients with hospital-acquired AKI.
  For patients that will not develop AKI during hospitalization, no other visits will be performed during the study, except for the discharge and follow-up visits.
Sampling Method: Probability Sample
Enrollment: 1456 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
90-day Mortality | 90 days
  Mortality at 90 days

SECONDARY OUTCOMES:
Phenotypes of acute kidney injury across geographic areas | Hospital stay (up to 90 days)
  Characteristics of acute kidney injury (clinical type and stage)
Staging of acute kidney injury across geographic areas | Hospital stay (up to 90 days)
  Characteristics of acute kidney injury (clinical type and stage)
Adherence to the International Club of Ascites recommendations for the management of AKI | Hospital stay (up to 90 days)
  Proportion of patients receiving treatment according to the International Club of Ascites recommmentations for the management of acute kidney injury
Progression of AKI | Hospital stay (up to 90 days)
  Progression of AKI will be defined as transition of AKI to a higher stage and/or need for RRT.
Resolution of AKI | Hospital stay (up to 90 days)
  Resolution of AKI will be defined as return of serum creatinine to a value within 0.3 mg/dl (26.5 mmol/L) of the baseline value. Partial response will be defined as regression of AKI to a lower stage with a reduction of serum creatinine to ≥0.3 mg/dl (26.5 mmol/L) above the baseline value
In-hospital mortality | Hospital stay (up to 90 days)
  Mortality during hospital stay
28-day mortality | 28 days
  Mortality at 28 days
Development of CKD | 90 days
  Chronic kidney disease will be defined as an estimated glomerular filtration rate <60 ml/min ml/min/1.73 m2 for >3 months. The Modification of Diet in Renal Disease equation will be used for estimating glomerular filtration rate

OTHER OUTCOMES:
Transfer to intensive care unit | Hospital stay (up to 90 days)
  Transfer to intensive care unit
Mechanical ventilation | Hospital stay (up to 90 days)
  Patients receiving mechanical ventilation
Renal replacement therapy | Hospital stay (up to 90 days)
  Patients receiving renal replacement therapy
Indication to RRT | Hospital stay (up to 90 days)
  Patients with indications to receive renal replacement therapy

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Piano, MD, Principal Investigator — Azienda Ospedaliera di Padova
Locations (38):
- United States (5):
  - Indiana University, Indianapolis, Indiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Baylor University Medical Center, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia
- Argentina (4):
  - Hospital de Gastroenterología "Dr. Carlos Bonorino Udaondo", Buenos Aires
  - Hospital Italiano, Buenos Aires
  - Hospital Nacional Prof. Alejandro Posadas, El Palomar
  - Universidad de Rosario, Rosario
- Hospital Federal de Bonsoccesso, Rio de Janeiro, Brazil
- Universidad de Chile, Santiago, Chile
- Shanghai Jiao Tong University School of Medicine, Shanghai, China
- Hvidovre Hospital, Copenhagen, Denmark
- Ain Shams University, Cairo, Egypt
- Black Lion Hospital, Addis Ababa, Ethiopia
- France (2):
  - Jean Minjoz University Hospital, Besançon
  - Hospital Beaujon, Clichy
- Germany (2):
  - University of Aachen, Aachen
  - University Hospital Munich, Munich
- Hospital of Debrecen, Debrecen, Hungary
- Institute of Liver and Biliary Sciences, New Delhi, India
- Italy (5):
  - IRCCS Azienda Ospedaliera-Universitaria di Bologna, Bologna
  - Università La Sapienza - Latina, Latina
  - Hospital Niguarda Milan, Milan
  - University and Hospital of Padua, Padua
  - Azienda Ospedaliero Universitaria Città della Salute e della Scienza di Torino, Torino
- Mexico (3):
  - Central Military Hospital, Mexico City
  - Hospital General, Mexico City
  - Instituto Nacional de Ciencias Médicas y Nutrición "Salvador Zubirán", Mexico City
- Erasmus Medical Center, Rotterdam, Netherlands
- Hospital de Clínicas Facultad de Ciencias Médicas U.N.A., Asunción, Paraguay
- Hospital Nacional D.A. Carrion, Lima, Peru
- Medical University of Warsaw, Warsaw, Poland
- University of Moscow, Moscow, Russia
- South Korea (2):
  - Hallym University Sacred Heart Hospital, Anyang
  - Hallym University College of Medicine, Chuncheon
- Spain (2):
  - Hospital Clinic, Barcelona
  - Hospital Vall D'Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Angeli P, Gines P, Wong F, Bernardi M, Boyer TD, Gerbes A, Moreau R, Jalan R, Sarin SK, Piano S, Moore K, Lee SS, Durand F, Salerno F, Caraceni P, Kim WR, Arroyo V, Garcia-Tsao G. Diagnosis and management of acute kidney injury in patients with cirrhosis: revised consensus recommendations of the International Club of Ascites. J Hepatol. 2015 Apr;62(4):968-74. doi: 10.1016/j.jhep.2014.12.029. Epub 2015 Jan 28. No abstract available. PMID 25638527
- [Derived] Patidar KR, Ma AT, Juanola A, Barone A, Incicco S, Kulkarni AV, Hernandez JLP, Wentworth B, Asrani SK, Alessandria C, Abdelkader NA, Wong YJ, Xie Q, Pyrsopoulos NT, Kim SE, Fouad Y, Torre A, Cerda E, Ferrer JD, Maiwall R, Simonetto DA, Papp M, Orman ES, Perricone G, Sole C, Lange CM, Farias AQ, Pereira G, Gadano A, Caraceni P, Thevenot T, Verma N, Kim JH, Vorobioff JD, Cordova-Gallardo J, Ivashkin V, Roblero JP, Maan R, Toledo C, Gioia S, Fassio E, Marino M, Nabilou P, Vargas V, Merli M, Goncalves LL, Rabinowich L, Krag A, Balcar L, Montes P, Mattos AZ, Bruns T, Mohammed A, Laleman W, Carrera E, Cabrera MC, Girala M, Samant H, Raevens S, Madaleno J, Kim RW, Arab JP, Presa J, Ferreira CN, Galante A, Allegretti AS, Takkenberg B, Marciano S, Sarin SK, Durand F, Gines P, Angeli P, Sola E, Piano S; International Club of Ascites GLOBAL AKI team. Global epidemiology of acute kidney injury in hospitalised patients with decompensated cirrhosis: the International Club of Ascites GLOBAL AKI prospective, multicentre, cohort study. Lancet Gastroenterol Hepatol. 2025 May;10(5):418-430. doi: 10.1016/S2468-1253(25)00006-8. Epub 2025 Mar 6. PMID 40058397